CLINICAL TRIAL: NCT02815865
Title: A Randomized Controlled Study Comparing Cervical Foley Catheter, Vaginal Dinoprostone and a Combination of the Two Methods for Induction of Labor
Brief Title: Comparing Cervical Foley Catheter, Dinoprostone and a Combination of the Two for Labor Induction
Acronym: Induction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Roni Levy, Head of labor and delivery, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12014kmc
Record Dates: First submitted 2016-02-26; First posted 2016-06-28 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Failed Medical or Unspecified Induction of Labor
Keywords: Primiparous; Foley catheter; Dinoprostone; Induction
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Foley catheter and pitocin (Active Comparator): Intervention: Foley catheter and pitocin Foley catheter will be inserted through the cervix and inflated with 80 ml saline, pitocin will be initiated 1 hour later in the delivery room
  Interventions: Device: Foley catheter and pitocin
- Foley catheter and dinoprostone (Active Comparator): Intervention: Foley catheter and dinoprostone Foley catheter will be inserted through the cervix and inflated with 80 ml saline dinoprostone 3 mg will be inserted 1 hour later to the posterior fornix
  Interventions: Device: Foley catheter and Dinoprostone
- Dinoprostone (Active Comparator): Intervention: Dinoprostone 3 mg will be inserted to the posterior fornix
  Interventions: Drug: Dinoprostone

INTERVENTIONS:
Device: Foley catheter and pitocin — Foley catheter will be inserted through the cervix and inflated with 80 ml saline, pitocin will be initiated 1 hour later in the delivery room
  Other Names: Ballon
  Arms: Foley catheter and pitocin
Device: Foley catheter and Dinoprostone — Foley catheter will be inserted through the cervix and inflated with 80 ml saline Dinoprostone 3 mg will be inserted 1 hour later to the posterior fornix
  Arms: Foley catheter and dinoprostone
Drug: Dinoprostone — Dinoprostone 3 mg will be inserted to the posterior fornix
  Arms: Dinoprostone

SUMMARY:
The investigators intend to conduct a randomized clinical trial comparing 3 methods of induction of labor in term primiparous women with singleton. First group will be women induced with Foley catheter and pitocin, second group Foley catheter and vaginal dinoprostone and third group will be induced with vaginal dinoprostone alone. The investigators compare time for induction to delivery and way of delivery.

DETAILED DESCRIPTION:
Introduction:

Labor induction, an iatrogenic initiation of labor is one of the most common obstetric procedures performed nowadays. The rate of induction of labor more than doubled from 1990 through 2010 from 9.6% to 23.8% in the United State alone. There are many methods to promote labor induction, including mechanical and pharmacological methods that can be used alone or in conjugation. Choosing the right method for the right patient can be challenging, and up until now there is limited information regarding the most suitable and effective approach for cervical ripening and labor induction. Out of the vast options for cervical ripening, the Foley catheter and vaginal prostaglandins are frequently used. To date, few clinical trials have compared the different methods to evaluate the effectiveness and the risk in each method. Two randomized controlled trials compared the Foley catheter method with the vaginal dinoprostone method. In one study, the Foley catheter was found to be superior to the vaginal dinoprostone with regards to time to delivery, whereas in the other study no difference was found. In an additional trial, Foley bulb with vaginal Misoprostol was compared to Misoprostol alone. The first treatment resulted in a shorter time to delivery. These finding did not correlate with previous trials that either found no difference or superiority to Misoprostol alone. A recent study comparing Foley catheter with PGE2 in term oligohydramnios pregnancies showed that time to delivery was shorter in the PGE2 group. A meta-analysis comparing Misoprostol with dinoprostone showed that the first is more effective, but the latter is safer. Since in some obstetrics conditions such as preeclampsia and Intrauterine growth restriction (IUGR) an expeditious induction of labor may be needed, a combination of methods may fasten the induction to delivery interval. A recent study presented as an oral presentation at the society of maternal fetal medicine a month ago used a combination of Foley catheter and prostaglandins to induce labor. They found that this arm had the shorter induction to delivery time and had no serious side effects.

In this study, The investigators intend to compare the mechanical (Foley catheter combined with Oxytocin) method, to a pharmacological one (dinoprostone-PGE2) and to a combination of the two methods in cervical ripening in an unfavorable cervix. The investigators will also examine if using the two methods in tandem will provide an additive effect.

The study will include 3 groups; in each group about 100 participants will be enrolled, which will be suited to the including and excluding criteria. The investigators have about 200 inductions per year of primigravida women. The investigators expect to enroll 300 participants in about 2 years' time.

On enrollment the patient will receive a number and will be assigned to one of the three groups. All the participants will be assigned to a 20 minute reassuring monitor before insertion the device.

A perineal US will be performed before the intervention to evaluate Angle of progression (AOP), cervical length and head position.

Group 1: Foley and Oxytocin protocol The patient will lie in a lithotomy position and will be covered by sterile sheets. A direct visualization of the cervix will be achieved with sterile speculum, the cervix will be sterilized with iodine, if the patient is allergic to iodine "septal- scrub" will be used. The Foley will be inserted through the internal cervical os, filled with 80 ml of normal saline, and taped to the patient thigh with gentle traction. An hour after placing the Foley bulb, monitor will be performed. If less than 3 contractions per 10 min interval appears in the monitor the patient will be transferred to the delivery room and Oxytocin will be administrated. If 3 contraction or more appear in 10 min. interval, further intervention will be personalized according to medical decision.

The Foley catheter will be removed if any of the following will occur:

1. Expulsion
2. Non reassuring fetal heart rate, NRFHR
3. Tachysystole
4. spontaneous rupture of membranes, SROM
5. If 24 12 hours elapsed since placement.

Group 2:

Foley with dinoprostone protocol. First the Foley bulb will be placed as instructed above. An hour after placing the Foley bulb, a monitor will be performed. If less than 3 contractions per 10 min. interval appears in the monitor a propess tape will be placed in the posterior fornix. The patient will be left recumbent for 30 minutes. One hour after placing the dinoprostone, fetal monitor will be performed. If less than 3 contractions per 10 min interval appears in the monitor the patient will be remained for observation and a monitor will be performed every 6 hours. If after placing the Foley bulb 3 contractions or more appear in 10 minutes interval the patient will be excluded from the research and further intervention will be personalized according to medical decision

Group 3 Dinoprostone protocol Dinoprostone will be removed from the freezer in direct connection with insertion. The patient will lie in a lithotomy position. Dinoprostone will be inserted to the posterior vaginal fornix using small amount of water soluble lubricant according to the manufactory protocol. The reminding of the tap will be inserted to the vagina. The patient will be left recumbent for 30 minutes. An hour after placing the dinoprostone, fetal monitor will be performed and then every 6 hours. If less than 3 contractions per 10 min interval appears in the monitor the patient will be transferred for observation and a monitor will be performed every 6 hours. If 3 contraction or more appear in 10 min. interval the patient will be examined and in dilatation of 3 cm or more will be transferred to the delivery room.

The dinoprostone will be removed if any of the following will occur:

1. NRFHR
2. Tachysystole
3. SROM
4. If 24 hours elapsed since placement In all the groups, if after 24 hours since the start of the study, the bishop score will be still less than 6 and active labor will not initiate the same method (study arm) will be repeated. If after the second try the cervix is still unripe the patient will be defined as failed induction.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women
* 37 weeks pregnant or more
* cephalic live singleton,
* intact membranes
* Unfavorable cervix (bishop's score 6 or less)

Exclusion Criteria:

* Previous cesarean section or other uterine surgery
* severe IUGR
* severe preeclampsia
* Fetal malpresentation
* Multiple gestation
* Spontaneous labor (3 contraction in 10 min)
* Premature rupture of membranes, PROM
* Category 2 or greater fetal heart rate tracing
* Contraindication for vaginal delivery
* Fever
* Vaginal bleeding (more than spotting or bloody show)
* Severe IUGR
* HIV carrier
* Sensitivity to either latex or PGE2
* polyhydramnios

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Time from induction to delivery (in hours) | up to 24 hours
Mode of delivery | up to 24 hours
  Vaginal delivery or Cesarean section

SECONDARY OUTCOMES:
Time form induction to active labor (in hours) | up to 24 hours
Rate of deliveries within 24 hours | up to 24 hours
Tachysystole | up to 24 hours
  monitor recording of 5 or more contraction in a 10 minutes period with fetal heart deceleration
Neonatal Apgar scores (in a 1-10 scale) | up to 24 hours
  Neonatal Apgar score in the first, 5th and 10th minutes after the delivery
Neonatal intensive care unit admission | up to 72 hours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Martin JA, Hamilton BE, Ventura SJ, Mathews TJ. Births: final data for 2010. Natl Vital Stat Rep 2012;61:1-72. 2. Jozwiak M, Oude Rengerink K, Ten Eikelder ML, van Pampus MG, Dijksterhuis MG, de Graaf IM, et al. Foley catheter or prostaglandin E2 inserts for induction of labour at term: an open-label randomized controlled trial (PROBAAT-P trial) and systematic review of literature. European journal of obstetrics, gynecology, and reproductive biology. 2013;170(1):137-45. 3. Carbone JF, Tuuli MG, Macones GA. Combination of Foley bulb and vaginal misoprostol compared with vaginal misoprostol alone for cervical ripening and labor induction: a randomized controlled trial. Obstetrics and gynecology. 2013;121(2 Pt 1):247-52. 4. Kashanian M, Akbarian AR, Fekrat M. Cervical ripening and induction of labor with intravaginal misoprostol and Foley catheter cervical traction. International journal of gynaecology and obstetrics: the official organ of the International Federation of Gynaecology and Obstetrics. 2006;92(1):79-80. 5. Chung JH, Huang WH, Nageotte MP. A prospective randomized controlled trial that compared misoprostol, Foley catheter, and combination misoprostol-Foley catheter for labor induction. AJOG. 2003;189(4):1031-5. 6. LD Levine, S. Parry. MA. Elovitz. Foley or Misoprostol for the Management of Induction (The 'FOR MOMI' trial): A four-arm randomized clinical trial. AJOG 214, 1, S4, 2016.
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264